CLINICAL TRIAL: NCT03038061
Title: Ultrasound Detection of Presence of Diaphragm in the Region of Lung Monitoring Using Electrical Impedance Tomography During Laparoscopic Surgery
Brief Title: Ultrasound Detection of Position of Diaphragm During Laparoscopic Surgery
Acronym: UDLaS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Czech Technical University in Prague (Other)
Collaborators: Military University Hospital, Prague (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: NVT108-8/104-2015/ÚVN
Record Dates: First submitted 2017-01-28; First posted 2017-01-31 (Estimated); Last update posted 2021-02-25 (Actual); Status verified 2021-02

CONDITIONS: Laparoscopy
Keywords: Diaphragm; EIT; Laparoscopy

STUDY DESIGN:
Intervention Model Description: Single group assignment. Approx. 20 patients during laparoscopic surgery with capnoperitoneum.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental group (Experimental): Patients undergoing Laparoscopic Surgery
  Interventions: Other: Patients undergoing Laparoscopic Surgery

INTERVENTIONS:
Other: Patients undergoing Laparoscopic Surgery — Data are to be obtained at three phases at supine horizontal position (during spontaneous breathing, at mechanically ventilated patient under general anesthesia with muscle relaxation and at mechanically ventilated patient under general anesthesia with muscle relaxation during insufflation of carbon dioxide into the peritoneal cavity to achieve exposure during laparoscopic surgery).

SUMMARY:
Position of diaphragm in the region of electrical impedance tomography measurement is to be determined by ultrasound in approx. 20 patients undergoing laparoscopic surgery. Data are to be obtained at three phases at supine horizontal position (during spontaneous breathing, at mechanically ventilated patient under general anesthesia with muscle relaxation and at mechanically ventilated patient under general anesthesia with muscle relaxation during insufflation of carbon dioxide into the peritoneal cavity to achieve exposure during laparoscopic surgery).

DETAILED DESCRIPTION:
During laparoscopic surgery, insufflation of carbon dioxide into the peritoneal cavity is conducted in order to optimize working space for surgeons. As a side effect, the abdominal pressure alters physiological thoraco-abdominal configuration and pushes the diaphragm and lungs cranially. Since lung image acquired by electrical impedance tomography (EIT) depends on the conditions within the thorax and abdomen, it is crucial to know the diaphragm position to analyze the effect of cranial shift of diaphragm on EIT images of the thorax. Presence of diaphragm in the region of EIT measurement is to be determined by ultrasound in approx. 20 patients undergoing laparoscopic surgery. Data are to be obtained at three phases at supine horizontal position (during spontaneous breathing, at mechanically ventilated patient under general anesthesia with muscle relaxation and at mechanically ventilated patient under general anesthesia with muscle relaxation during insufflation of carbon dioxide into the peritoneal cavity to achieve exposure during laparoscopic surgery). The results of this study will serve during design of a subsequent study dealing with optimization of EIT electrode belt position during laparoscopic surgery.

ELIGIBILITY:
Inclusion Criteria:

- patients undergoing abdominal laparoscopic surgery

Exclusion Criteria:

* morbid obesity
* standard exclusion criteria for electrical impedance tomography according to the manufacturer

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2015-12-01 (Actual); Primary Completion 2021-02-24 (Actual); Study Completion 2021-02-24 (Actual)

PRIMARY OUTCOMES:
Position of Diaphragm Detected by Ultrasound | Within one laparoscopic surgery (1-3 hours)
  Measurement in midclavicular line

CONTACTS AND LOCATIONS:
Overall Officials: Karel Roubik, Prof. Ph.D., Study Director — Czech Technical University in Prague; Martin Müller, Principal Investigator — Czech Technical University in Prague / Military University Hospital, Prague
Locations (1):
- Military University Hospital, Prague, Czechia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Valenza F, Chevallard G, Fossali T, Salice V, Pizzocri M, Gattinoni L. Management of mechanical ventilation during laparoscopic surgery. Best Pract Res Clin Anaesthesiol. 2010 Jun;24(2):227-41. doi: 10.1016/j.bpa.2010.02.002. PMID 20608559
- [Background] Staehr-Rye AK, Rasmussen LS, Rosenberg J, Steen-Hansen C, Nielsen TF, Rosenstock CV, Clausen HV, Sorensen MK, VON H Regeur J, Gatke MR. Minimal impairment in pulmonary function following laparoscopic surgery. Acta Anaesthesiol Scand. 2014 Feb;58(2):198-205. doi: 10.1111/aas.12254. Epub 2014 Jan 2. PMID 24383568
- [Derived] Buzkova K, Muller M, Rara A, Roubik K, Tyll T. Ultrasound detection of diaphragm position in the region for lung monitoring by electrical impedance tomography during laparoscopy. Biomed Pap Med Fac Univ Palacky Olomouc Czech Repub. 2018 Mar;162(1):43-46. doi: 10.5507/bp.2018.005. Epub 2018 Feb 21. PMID 29467544
- Available data/document: Informed Consent Form — http://ventilation.fbmi.cvut.cz/wp-content/uploads/2017/01/Informed-Consent-Form.pdf — Informed Consent